CLINICAL TRIAL: NCT03323762
Title: Effect of Remote Ischemic Conditioning on Blood Pressure and Inflammatory Response in Women With Pre-eclampsia and Gestational Hypertension
Brief Title: Effect of RIC on BP and Inflammatory Response in Women With Pre-eclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Randers Regional Hospital (Other); Herning Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIC & pre-eclampsia
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2019-01

CONDITIONS: Pre-Eclampsia; Mild; Gestational Hypertension
Keywords: Pre-Eclampsia; Mild; Pre-Eclampsia; Moderate; Gestational Hypertension; Remote ischemic conditioning
MeSH Terms: conditions — Pre-Eclampsia; Lymphoma, Follicular; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RIC (Experimental): RIC treatment arm The CellAegis auto RIC (automated blood pressure cuff) will be placed on the upper arm and inflated to 200 mmHg for 5 minutes followed by 5 minutes of deflation. The programmed cycle is repeated 4 times in total, summing up to a total treatment length of 35 minutes.
  The treatment will be carried out on the morning of day 2 to day 7 by the participants themselves at their home.
  Interventions: Device: Remote Ischaemic Conditioning (RIC)

INTERVENTIONS:
Device: Remote Ischaemic Conditioning (RIC) — The CellAegis auto RIC (automated blood pressure cuff) will be placed on the upper arm and inflated to 200 mmHg for 5 minutes followed by 5 minutes of deflation. The programmed cycle is repeated 4 times in total, summing up to a total treatment length of 35 minutes

SUMMARY:
The aim of this pilot cohort study is to investigate whether treatment with remote ischemic conditioning (RIC) has a beneficial effect on blood pressure as well as the immune system in pregnant women with newly diagnosed hypertension (> 140/58 mm Hg) or pre-eclampsia before gestational week 37+3.

DETAILED DESCRIPTION:
Pre-eclampsia, which affects about 2 to 7% of pregnancies, is a major cause of maternal and perinatal morbidity and mortality.

The onset of clinical symptoms (hypertension, proteinuria or end- organ dysfunction), are often seen in the last trimester of a pregnancy.

The disease can have major consequences for both the child and the mother. Yet there are only very limited treatment options, where induced labour is the only healing treatment. Today, the treatment consists in limiting blood pressure increase with medical treatment, whereby the pregnancy most often can result in term delivery.

Remote Ischaemic Conditioning (RIC) achieved by an automatic inflation of a blood pressure cuff to induce four 5-minute cycles of limb ischaemia and reperfusion, is a treatment that has been found to decrease the inflammatory response and lower blood pressure in states of myocardial infarction, chronic heart failure, and stroke.

The treatment is virtually a cost-free non-pharmacological and non-invasive therapeutic strategy performed by the patient herself in her home.

However, whether RIC actually can improve clinical outcomes in relation to lowering blood pressure and the inflammatory response in pregnant women with newly diagnosed hypertension is yet to be investigated.

Aim and endpoint:

The aim of this pilot cohort study is to investigate whether treatment with remote ischemic conditioning (RIC) has a beneficial effect on blood pressure as well as the immune system in pregnant women with newly diagnosed hypertension (> 140/58mm Hg) or pre-eclampsia before gestational week 37+3.

Primary end-point • Median arterial blood pressure after 6 days of treatment

Secondary end-point

• Changes in the inflammatory response

Design and method:

In a pilot cohort study at Aarhus University Hospital, Regional Hospital Randers and Region Hospital Herning 20 pregnant women with signs of gestational hypertension or pre-eclampsia (systolic blood pressure above 140 and / or diastolic blood pressure over 85; +/- proteinuria, +/- clinical signs or subjective symptoms and signs) are to be enrolled.

The study flowchart:

Newly hospital referred women with signs of gestational hypertension or pre-eclampsia will be asked to participate. Informed consent will be obtained and blood pressure, blood samples, and weight will be measured.

* Day 1: resting day at home - blood pressure measuring
* Day 2-7: Morning: Blood pressure measuring and RIC treatment. Evening: blood pressure measuring
* Day 7: In hospital: Blood samples and weight will be measured.

Pros and cons:

In relation to the inflation of the blood pressure cuff temporary moderate pains in the treated arm might occur. Otherwise, the RIC is without side effects. Two extra blood samples of app. 50 ml each will be drawn, with a small risk of local infection exist.

The usefulness of the study The study is designed as a small pilot study. In which the set up will be tested and the effects on blood pressure and the inflammatory response in a relative small size will be explored. A larger randomised study will follow if the results show a positive trend.

Positive as well as negative and inconclusive results will be widely disseminated through national and international scientific journals and conferences.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure above 140 and/or
* Diastolic blood pressure above 85
* Proteinuria +/-
* Clinical signs / symptoms +/-

Clinical signs and symptoms of pre-eclampsia +/-

Exclusion Criteria:

• Eclampsia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Obs pre-eclampsia
Enrollment: 10 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Median arterial blood pressure | after 6 days of treatment
  Median arterial blood pressure after 6 days of treatment

SECONDARY OUTCOMES:
The inflammatory response | after 6 days of treatment
  Changes in the inflammatory response after 6 days of treatment
Medication | After 6 days of treatment
  prescription of antihypertensive

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Kristine Møller Liendgaard, Phd, MHSc., Principal Investigator — Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Aarhus University hospital, Aarhus
  - Herning Hospital, Herning
  - Randers Hospital, Randers

IPD SHARING:
Plan to Share IPD: No